CLINICAL TRIAL: NCT00466700
Title: Genotypes of Helicobacter Pylori in West African Children and Adults: Part 1: The Development and Evaluation of Minimally Invasive Techniques for Obtaining H. Pylori Isolates From Adults and Children in The Gambia
Brief Title: Helicobacter in The Gambia (Part 1)
Status: Completed | Type: Observational
Sponsor: Medical Research Council Unit, The Gambia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 06-0053
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Helicobacter Pylori
Keywords: Helicobacter pylori, Gambia, endoscopy, Africa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
H. pylori infection causes the stomach to become inflamed. The problem usually begins in childhood and leads to stomach problems in adult life. Study participants will be residents of The Gambia, West Africa, and will be studied at the Medical Research Council of Great Britain facility in Fajara, The Gambia. Up to 75 adults 18 years and older and 20 malnourished children 6 months to 2 years of age, who are undergoing endoscopy as part of their medical care, will be studied. (Endoscopy is when a thin, lighted device is used to look inside the body.) During this study procedure, tiny pieces of tissue, called biopsies, will be taken from the stomach and checked for H. pylori infection. Participants found to be infected will be given antibiotic treatment. Participation in the study will last approximately 72 hours.

DETAILED DESCRIPTION:
The overall goal in this pilot project is to implement and evaluate a new method for isolating Helicobacter pylori (H. pylori) strains from young children, and to compare these isolates with those obtained from adults from the same population. This is part I of the study, and part II is described in the Division of Microbiology and Infectious Diseases protocol 06-0004. The transition from childhood colonization to adult disease state may be affected by multiple factors including evolution of genotypes of colonizing H. pylori strains themselves, driven in part by the host response to infection. The hypothesis is that H. pylori strains from Gambian children will differ genetically from the strains of chronically colonized adults from the same community. Genetic and phenotypic characterization of pediatric and adult H. pylori isolates will test for fundamental differences between strains circulating in these 2 age groups, and thereby help evaluate the importance of strain selection and/or genome evolution in such high risk societies. Specific objectives are: to compare the range of genotypes obtained from H. pylori cultured from gastric biopsies from Gambian adults and children undergoing diagnostic upper endoscopy, with those obtained by culture of gastric juice aspirates from the same subjects. This will allow interpretation of results obtained from culture of nasogastric aspirates from children who do not require diagnostic endoscopy, when compared to gastric biopsy-derived H. pylori isolates. Most genotyping will entail polymerase chain reaction tests for virulence markers, limited (focused) DNA sequencing, and tests for susceptibility to metronidazole and frequency of forward mutation. The study population will consist of residents of The Gambia, West Africa. Up to seventy five adults of both sexes and all ages, who are undergoing diagnostic endoscopy as part of their clinical management, and 20 malnourished children of both sexes and less than 2 years of age, who are undergoing diagnostic endoscopy as part of their clinical management, will be studied. All subjects will be studied at the Medical Research Council of Great Britain research laboratories and clinical facility in Fajara, The Gambia. The main outcome measure will be the degree of relatedness between bacterial isolates. This will be assessed by visual comparison between random amplification of polymorphic DNA (RAPD) results, by comparison of genotype for alleles of interest, and definitively by sequencing of housekeeping genes to construct phylogenetic trees of relatedness, using the STAR program (a computer program for putting DNA sequences together for analysis) and multiple locus sequence typing (MLST) database. There are no outcome measures for human subjects. All laboratory investigations will be conducted upon bacterial isolates.

ELIGIBILITY:
Inclusion Criteria:

Adult Subjects: All consenting subjects referred for diagnostic upper endoscopy to the Medical Research Council (MRC) unit in Fajara will be eligible for inclusion, provided none of the exclusion criteria apply. In The Gambia, subjects aged 18 years and above are considered as adult. Subjects will be sampled only once.

Child Subjects: All subjects under 2 years of age referred for diagnostic upper endoscopy to the MRC unit in Fajara will be eligible for inclusion, provided their parents give informed consent and that none of the exclusion criteria apply. The minimum cut-off age for this study will be 6 months.

Exclusion Criteria:

Adult Subjects: Any contraindication to endoscopy and biopsy, such as as liver dysfunction, history of bleeding, history of other serious organ disease (for example, kidney, heart, lung), bleeding time prolonged to over 10 minutes, or unexpected findings such as esophageal or gastric stricture that limits endoscopic examination will exclude subjects from the study, as will the use of antibiotics during the previous 2 weeks. Specific tests such as bleeding times will be performed at the discretion of the supervising clinician, who is undertaking the diagnostic endoscopy for the subject's clinical benefit. In addition, if the endoscopist feels that prolonging the procedure by 2 or 3 minutes in order to take the research biopsies would not be advisable for any reason, the subject will be excluded from the study.

Child Subjects: Any contraindication to endoscopy and biopsy, such as as liver dysfunction, history of bleeding, history of other serious organ disease (for example, kidney, heart, lung), bleeding time prolonged to over 10 minutes, or unexpected findings such as esophageal stricture that limits endoscopic examination will exclude subjects from the study, as will the use of antibiotics during the previous 2 weeks. In addition, if the endoscopist feels that prolonging the procedure by 2 or 3 minutes in order to take the research biopsies would not be advisable for any reason, the subject will be excluded from the study. Specific tests such as bleeding times will be performed at the discretion of the supervising clinician, who is undertaking the diagnostic endoscopy for the subject's clinical benefit.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of rural subsistence farmers and semi-urban dwellers attending the clinic at the MRC research laboratories in Fajara, The Gambia. The study will be comprised of subjects who are undergoing endoscopy for diagnostic purposes within the endoscopy unit at Fajara.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The degree of relatedness between bacterial isolates | 4 years
  This will be assessed by visual comparison between RAPD results, by comparison of genotypes for alleles of interest, and definitively by sequencing of housekeeping genes to construct phylogenetic trees of relatedness, using the STAR program (a computer program for putting DNA sequences together for analysis) and MLST database.
  There are no outcome measures for human subjects. All laboratory investigations will be conducted upon bacterial isolates There are no outcome measures for human subjects. All laboratory investigations will be conducted upon bacterial isolates

CONTACTS AND LOCATIONS:
Overall Officials: Richard Adegbola, PhD, FRCPath, Principal Investigator — Medical Research Council Unit, The Gambia
Locations (1):
- Medical Research Council's Laboratories, Banjul, The Gambia